CLINICAL TRIAL: NCT02980627
Title: iOmit: Reducing Intentional Insulin Misuse in Type 1 Diabetes
Acronym: iOmit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00068040; 1R21DK106603-01A1 (NIH)
Record Dates: First submitted 2016-07-08; First posted 2016-12-02 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes Mellitus; Eating Disorders
Keywords: Eating Disorders; Diabulimia; ED-T1DM; Type 1 Diabetes; Mobile Technology; Acceptance and Commitment Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders; Diabulimia | interventions — Therapeutics; Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy with Mobile App Enhancement (Experimental): Participants will complete initial assessments and then take part in a 3-month intervention consisting of 12 weekly individual therapy sessions with daily RR app use between sessions. At the end of the 3-month intervention period, an exit interview will be conducted and participants will complete a second assessment consisting of questionnaires and an ED diagnostic interview, a blood specimen for HbA1c, and 3-days of blinded CGM monitoring. Participants will then enter a 6-month follow-up period during which time they may continue to use the app, but will no longer attend individual sessions. Participants will be return to the clinic at 6 and 9 months for follow-up.
  Interventions: Behavioral: Therapy with Mobile App Enhancement

INTERVENTIONS:
Behavioral: Therapy with Mobile App Enhancement — Treatment includes 12 weekly therapy sessions with daily RR app use between sessions. Intervention is CBT-based and specifically draws from ACT. ACT is a contextual behavior therapy that emphasizes the function of behavior (e.g., affect regulation) and helps individuals accept (or "tolerate") emotional discomfort for a broader purpose (i.e., personal values). Broadly, treatment will focus on improving diabetes management by increasing patients' capacity to effectively cope with psychological barriers to self-care using acceptance and mindfulness strategies.
  Other Names: Recovery Record; Acceptance and Commitment Therapy; ACT; Mobile Technology

SUMMARY:
Individuals with type 1 diabetes who intentionally omit insulin to lose weight are at high risk for diabetes-related medical complications and premature death. Conventional eating disorder (ED) treatments are not as effective for these patients, suggesting that they need a more tailored treatment approach and one that includes intervention at the time and place when they are making decisions about their diabetes self-management. The goal of treatment development project is to modify an existing mobile application (app) for EDs (Recovery Record; RR) to address the unique needs of adults with type 1 diabetes (T1D) who intentionally omit their insulin for weight control, and test whether app-supported individual treatment decreases eating disorder (ED) symptoms and improves metabolic control. The investigator will also gather preliminary data on the impact of the intervention on health care utilization and costs and calculate attrition to assess feasibility.

The investigators hypothesize that (1) participants will evidence significant decreases in mean blood glucose, (2) participation in routine medical care will increase and emergency visits will decrease, (3) the percentage of time participants are hyperglycemic will decrease, (4) participant scores on the DEPS-R will decrease and (5) participant scores on the EDE will decrease.

DETAILED DESCRIPTION:
Intentional insulin omission for weight control is a significant problem in the clinical management of type 1 diabetes (T1D); despite this, there are no effective treatments. Combining the use of mobile technology with individual therapy may help individuals with T1D identify their triggers for insulin omission in their natural environment and cope more effectively. In the current study, the investigators examine whether pairing a mobile application, Recovery Record, with individual therapy helps reduce intentional insulin omission for weight control among individuals with T1D. In Phase 1, the investigators build T1D-specific content into the Recovery Record app based on our empirical evidence of triggers for insulin omission and qualitative feedback from T1D patients. The fully functional app is beta tested with 10 T1D patients who intentionally omit insulin. In Phase 2, 25 T1D patients that misuse insulin complete 3 months of app-supported individual treatment and 6 months of follow-up. The investigators test whether treatment is associated with decreases in mean blood glucose, eating disorder symptoms and emergency care utilization. The investigators also test whether frequency of app use in months 0-3 corresponds with outcomes, and calculate attrition..

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 or older
2. Diagnosed with T1D
3. Positive for insulin misuse for weight control
4. HbA1c ≥ 7.5
5. Approved for participation by their physician
6. Agrees to continue care with their current physician with consent to contact
7. Access to a Smartphone

Exclusion Criteria:

1. Non-English speaking
2. Cognitive impairments that preclude independent management of T1D

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Metabolic Control (Change in HbA1c) | Baseline, 3-months, 6-months and 9-months

SECONDARY OUTCOMES:
Mobile Technology Engagement (Frequency of Use) | Daily monitoring for 3 months
  Improvements in metabolic control will correspond with treatment engagement as reflected in frequency of app use from 0-3 months
Adequate Insulin Dosing (Frequency) | Baseline, 3-months, 6-months and 9-months
  Participants will report less frequent under-dosing of insulin
Medical Utilization: Total Number of Primary Care Visits | Baseline, 3-months, 6-months, and 9-months
Medical Utilization: Total Number of Emergency Department Care Visits | Baseline, 3-months, 6-months, and 9-months
Participant Engagement in Treatment as evidenced by attendance/treatment completion | 3 months
  Attrition will be < 20%
Improvement in Metabolic Control; CGM Continuous Glucose Monitoring | Baseline, 3-months
Decrease in Diabetes-Specific Eating Disorder symptomatology | Baseline, 3-months, 6-months, and 9-months
Decrease in Overall Eating Disorder symptomatology | Baseline, 3-months, 6-months, and 9-months

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Merwin, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Health System, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merwin RM, Dmitrieva NO, Honeycutt LK, Moskovich AA, Lane JD, Zucker NL, Surwit RS, Feinglos M, Kuo J. Momentary Predictors of Insulin Restriction Among Adults With Type 1 Diabetes and Eating Disorder Symptomatology. Diabetes Care. 2015 Nov;38(11):2025-32. doi: 10.2337/dc15-0753. Epub 2015 Sep 17. PMID 26384389
- [Background] Merwin RM, Moskovich AA, Dmitrieva NO, Pieper CF, Honeycutt LK, Zucker NL, Surwit RS, Buhi L. Disinhibited eating and weight-related insulin mismanagement among individuals with type 1 diabetes. Appetite. 2014 Oct;81:123-30. doi: 10.1016/j.appet.2014.05.028. Epub 2014 May 29. PMID 24882448
- [Derived] Merwin RM, Moskovich AA, Babyak M, Feinglos M, Honeycutt LK, Mooney J, Freeman SP, Batchelder H, Sangvai D. An open trial of app-assisted acceptance and commitment therapy (iACT) for eating disorders in type 1 diabetes. J Eat Disord. 2021 Jan 6;9(1):6. doi: 10.1186/s40337-020-00357-6. PMID 33407910
- See also: Acceptance and Commitment Therapy at Duke University Medical Center — http://www.ACTatDuke.org